CLINICAL TRIAL: NCT07053267
Title: Effects of Acute Consumption of Ice Cream Enriched With Cimarron Bean Extruded on Metabolic Responses in Adults: A Non-Randomized Clinical Trial
Brief Title: Acute Postprandial Effects of Functional Ice Cream With Cimarrón Bean Extrudate in Adults
Acronym: ICE-CBE-GLULIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Talca (Other)
Collaborators: Centro de Estudios en Alimentos Procesados (Other)
Responsible Party: Principal Investigator, Iván Palomo González, Principal Investigator, University of Talca
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ACU-HEP-UTALCA-F29-2021
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Disease Risk Factor; Insulin Resistance; Overweight (BMI > 25); Hyperglycaemia
Keywords: Phaseolus vulgaris; Ice cream; Postprandial metabolism; Functional food; Dietary intervention; Glucose response; Insulin response; Lipid profile
MeSH Terms: conditions — Insulin Resistance; Overweight; Hyperglycemia

STUDY DESIGN:
Intervention Model Description: This is a parallel-group clinical trial in which participants were non-randomly assigned to one of two arms: a single-dose intervention group consuming a functional ice cream enriched with Cimarrón bean extrudate, or a placebo group consuming an identical ice cream without the functional ingredient. Both groups were assessed in parallel for postprandial metabolic responses after a single intervention day.
Who Masked: Participant
Masking Description: Participants were blinded to the intervention type (placebo vs. functional ice cream) by providing both ice creams with identical appearance, texture, and flavor.
  The investigators were not blinded due to the need to manage logistics and sample handling. However, participants were unaware of their group assignment to minimize bias in self-reported adherence and perception of effects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Ice Cream with Cimarrón Bean Extrudate (Experimental): Participants consume a single 100 g portion of ice cream enriched with 10 g Cimarrón bean extrudate.
  Interventions: Dietary Supplement: Funrional Ice Cream
- Placebo Ice Cream (Placebo Comparator): Participants consume a single 100 g portion of placebo ice cream identical in appearance and flavor, but without the Cimarrón bean extrudate.
  Interventions: Dietary Supplement: Placebo Ice Cream

INTERVENTIONS:
Dietary Supplement: Funrional Ice Cream — Single 100 g serving of ice cream enriched with 10 g of Cimarrón bean extrudate, administered after an overnight fast to evaluate postprandial metabolic responses.
  Arms: Functional Ice Cream with Cimarrón Bean Extrudate
Dietary Supplement: Placebo Ice Cream — Single 100 g serving of placebo ice cream identical in flavor, texture, and appearance, but without Cimarrón bean extrudate, administered after an overnight fast to evaluate postprandial metabolic responses.
  Arms: Placebo Ice Cream

SUMMARY:
The goal of this non-randomized clinical trial is to evaluate the acute postprandial metabolic effects of a functional ice cream enriched with Cimarrón bean (Phaseolus vulgaris L. local variety Cimarrón) extrudate in adults with at least one cardiovascular risk factor.

The main questions it aims to answer are:

* Does the functional ice cream reduce postprandial glucose and insulin levels?
* Does it affect postprandial lipid concentrations?

Researchers will compare participants receiving a single dose of the functional ice cream containing 10 g of extrudate per 100 g to placebo version without extrudate, both ice creams are identical in appearance and taste.

Participants will:

* Attend a clinical visit in fasting conditions (10-12 hours).
* Provide baseline blood samples for glucose, insulin, and lipid profile.
* Consume a single 100 g portion of functional or placebo ice cream.
* Provide postprandial blood samples at defined time points.

DETAILED DESCRIPTION:
This Study trial is to evaluate the acute postprandial metabolic effects of a functional ice cream with Cimarrón bean (Phaseolus vulgaris L. local variety Cimarrón) extrudate in adults with at least one cardiovascular risk factor.

It is a non-randomized, single-blind, parallel-group clinical trial with two arms: intervention (functional ice cream) and control (placebo ice cream). Both products are matched for texture, flavor, and appearance to maintain participant blinding.

Participants arrive at the clinic after a 10-12 hour fast. Baseline blood samples are collected for glucose, insulin, and lipid profile. They then consume one 100 g portion of the assigned ice cream. Blood samples are collected postprandially at 120 minutes to assess changes in glucose, insulin and lipid profile.

The study aims to determine whether the functional ice cream modifies postprandial glycemic and lipemic responses, providing insight into its potential use as a dietary strategy to reduce cardiometabolic risk.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participant
* Men and women aged 20-59 years
* Willingness to participate and provide written informed consent

Exclusion Criteria:

* Documented food allergies, especially to legumes or beans
* Diagnosed liver, kidney, autoimmune diseases or severe illnesses such as cancer.
* Diagnosed gastrointestinal diseases including inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis), celiac disease, or any condition causing chronic gastrointestinal symptoms such as malabsorption, persistent diarrhea, or gastrointestinal bleeding

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Postprandial Glucose Concentration | Baseline and 120 minutes after consumption
  Blood glucose levels will be measured at fasting (baseline) and at 120 minutes following the intake of either functional or placebo ice cream. Outcome will be expressed in mg/dL.
Change in Postprandial Insulin Concentration | Baseline and 120 minutes after consumption
  Blood insulin levels will be assessed at fasting and at 120 minutes post-consumption. Outcome will be expressed in µIU/mL.

SECONDARY OUTCOMES:
Change in Postprandial Lipid Profile | Baseline and 120 minutes after consumption.
  Total cholesterol, HDL-c, LDL-c, and triglycerides will be measured at baseline and at 120 minutes post-consumption. Values will be expressed in mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan F Palomo González, PhD. Biomedical Science, Principal Investigator — University of Talca; Eduardo J Fuentes Quinteros, PhD. Science research, Principal Investigator — University of Talca
Locations (1):
- Universidad de Talca, Talca, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: Undecided
The plan to share individual participant data (IPD) has not yet been determined. The decision will depend on future publication plans, data management policies, and ethical considerations regarding participant privacy.